CLINICAL TRIAL: NCT05377125
Title: Neural Mechanisms of Response Inhibition Training for Obsessive-Compulsive Disorder and Related Conditions
Brief Title: Neural Mechanisms of Response Inhibition Training for OCRD
Acronym: OCRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00042324
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder; Tricholemmoma; Skin-Picking
Keywords: OCD; Trichotillomania; Excoriation; Response Inhibition
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Excoriation Disorder; Trichotillomania

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the two training groups in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed which of the two training conditions they are assigned to. Independent outcome (IE) evaluator will remain blinded to the assigned condition of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Response Inhibition Training (RIT) (Experimental): Response Inhibition Training (RIT) is a about 40-level computer game designed to offer systematic practice of RI. Participants use the computer keyboard and mouse to respond to the demands of trials that are designed to offer training on response inhibition abilities, including suppressing pre-potent but irrelevant stimuli and responses. Each training session will last approximately 45 minutes. All participants will be offered a minimum of 8 sessions. Throughout training, we will continually monitor their behavioral RI index (= stop signal reaction time; SSRT) using a stop-signal task. If a participant's Index SSRT fails to reach a criterion-level reduction (i.e., approximately 1 SD) after the standard 8 session intervention, the RIT intervention will be extended up to 16 sessions until the criterion-level improvement in behavioral RI is attained.
  Interventions: Behavioral: Computerized cognitive training
- Placebo Training (PLT) (Placebo Comparator): This training condition is designed to serve as an appropriate control condition for RIT, by providing no active ingredient of RI training components, while maintaining the overall training materials and structure similar. Similar to RIT, PLT uses the same task materials and a similar 40-level game structure. However, PLT will present simple RI-irrelevant visual judgment tasks to avoid changing RI-relate processes. The number of 45-min training sessions will be determined by their counterpart RIT participants through a yoked-control design.
  Interventions: Behavioral: Computerized placebo training

INTERVENTIONS:
Behavioral: Computerized cognitive training — This intervention offers 45-minute computerized training sessions to each participant. This intervention aims to improve the individual's RI capabilities. All participants will receive 8 to 16 sessions after being randomized to this condition.
  Arms: Response Inhibition Training (RIT)
Behavioral: Computerized placebo training — This intervention offers 45-minute computerized placebo cognitive training sessions to each participant. This intervention aims to exert no focused training on RI capabilities. All participants will receive 8 to 16 sessions after being randomized to this condition.
  Arms: Placebo Training (PLT)

SUMMARY:
The impaired ability to suppress an inappropriate but pre-potent response (response inhibition; RI) characterizes several debilitating clinical problems, including obsessive-compulsive and related disorders (OCRD) such as obsessive-compulsive disorder, trichotillomania, and skin picking disorder. There is a critical need to develop an effective and durable treatment for OCRDs with demonstrable evidence for improving impaired RI. The purpose of our project is to examine the impact of a novel computerized intervention, response inhibition training (RIT), on neural indices of RI, and examine the mechanistic link between engagement of the neural RI targets and change in OCRD symptoms. To this end, this project will conduct a randomized clinical trial for individuals with OCD, trichotillomania, and/or skin picking disorders. Participants will be randomly assigned to 8 to 16 sessions of computerized RIT or a computerized placebo training. Various clinical, behavioral, and brain-imaging data will be acquired to evaluate the training effects at baseline, post-training, and 1-month follow-up periods.

DETAILED DESCRIPTION:
Research has documented abnormal inhibition-related brain activity as well as impaired behavioral performance of RI in OCRD. Despite the growing evidence suggesting a RI deficit as a fundamental process in OCRD, no validated treatment exists that can directly alter RI deficits and in turn ameliorate OCRD symptoms. It is vital to develop a highly specific intervention that precisely engages a theoretically and empirically well-grounded target such as RI deficits, to significantly improve the efficacy of our intervention efforts. The overarching goal of this study is to examine whether the computerized cognitive training program can improve the neural indicators of the ability to inhibit inappropriate responses, and produce a clinically meaningful level of reduction in obsessive-compulsive disorder and related symptoms. Our central hypothesis is that cognitive training designed to enhance RI will improve neural indices: fronto-basal ganglia circuitry, especially right inferior frontal cortex of RI among individuals with OCRDs. We also hypothesize that the change in the RI neural circuit will mediate the consequent clinical improvements in OCRD symptomatology.

Phase I (R61) will aim to examine change in neural RI indices via the RIT intervention, Adults diagnosed with OCRD problems (OCD, TTM, or SPD) will be randomly assigned to the RIT or placebo control (PLT) condition. At pre- and post-training, neurobehavioral measures of RI will be taken, including the Stop-Signal Task (SST) assessing SSRT and fMRI task assessing rIFC activation. Each RIT participant will continue with the training within the range of 8 to 16 sessions until the criterion-level change in SSRT is attained (based on the ongoing SSRT estimation), with the PLT group receiving comparable levels of training. We will also collect 1-month follow-up data on functional outcomes in order to obtain information on the effect of the intervention on the OCRD symptom indices.

Phase II (R33) is identical to Phase I in the overall study procedures. Adults diagnosed with OCRD problems will be assigned to RIT or PLT. Analytic focus will be on the reduction in OCRD symptoms and their potential mediational pathway (rather than the change in the neural RI indices, which is the primary analytic focus in Phase I). Other than these differences, the overall flow and procedures of the study will be identical between Phases I and II.

The key assessments will include the fMRI tasks of the RI processes and clinician-administered measures of OCRD symptoms. There are other self-reported, computerized, and clinician-administered measures that will be administered across various points over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60
* moderate level of OCRD symptoms (Yale-Brown Obsessive Compulsive Scale total ≥ 16, Massachusetts General Hospital-Hair pulling Scale total ≥ 12, or Skin Picking Scale-Revised total ≥ 7)
* a primary diagnosis of OCRD (i.e., OCD, TTM, or SPD)
* estimated IQ > 80
* presence of a RI deficits (SSRT ≥ 215ms).

Exclusion Criteria:

* Current substance use disorder
* Severe ADHD
* Lifetime diagnosis of psychotic disorder, bipolar disorder, or schizophrenia
* Current psychotherapy
* Change in psychotropic medication status within 8 weeks before the study or during the study
* Use of stimulant medication
* Active suicidal risk
* Contraindications for MRI procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in obsessive-compulsive disorder symptom severity over time | Week 0, Week 4, Week 8 ~ 12
  Depending on participant's primary diagnostic condition, Yale-Brown Obsessive Compulsive Scale (YBOCS) will be used as the primary outcome measure for assessing the change in OCD symptoms over time.
  The total score ranges between 0 and 40 with higher scores indicating worse outcomes (= more severe symptoms).
Change in compulsive hair pulling symptom severity over time | Week 0, Week 4, Week 8 ~ 12
  Depending on participant's primary diagnostic condition, National Institute of Mental Health - Trichotillomania Symptom Severity Scale (NIMH-TSS) will be used as the primary outcome measure for assessing the change in hair pulling symptoms over time.
  The total score ranges between 0 and 25 with higher scores indicating worse outcomes (= more severe symptoms).
Change in compulsive skin picking symptom severity over time | Week 0, Week 4, Week 8 ~ 12
  Depending on participant's primary diagnostic condition, Yale-Brown Obsessive Compulsive Scale modified for Neurotic Excoriation (NE-YBOCS) will be used as the primary outcome measure for assessing the change in skin picking symptoms over time.
  The total score ranges between 0 and 40 with higher scores indicating worse outcomes (= more severe symptoms).
Change in activation in the right inferior frontal cortex (rIFC) | Week 0, Week 4
  Change in the level of blood-oxygen-level-dependent (BOLD) signal activation in the right inferior frontal cortex (rIFC) will be assessed using the stop-signal task (SST) that will be administered while the participant undergoes a functional magnetic resonance imaging procedure.

SECONDARY OUTCOMES:
Change in the Clinical Global Impression Scale | Week 0, Week 4, Week 8 ~ 12
  The Clinical Global Impression Scale (CGI-I) is a clinician-administered rating scale on the overall improvement of the participant's condition throughout treatment.
  The rating score ranges between 1 and 8 with higher scores indicating worse outcomes (= more severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Hanjoo Lee, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee; Christine Larson, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- UWM Anxiety Disorders Laboratory, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No